CLINICAL TRIAL: NCT01778413
Title: Virological and Immunological Safety of a Dose Reduction Strategy Antiretroviral Regimen With Efavirenz / Tenofovir / Emtricitabine
Acronym: A-TRI-WEEK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anna Cruceta (Other)
Responsible Party: Sponsor-Investigator, Anna Cruceta, Project manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-TRI-WEEK
Record Dates: First submitted 2013-01-18; First posted 2013-01-29 (Estimated); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: HIV
MeSH Terms: interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATRIPLA three times a week. (Experimental): Atripla (600 mg/200 mg/245 mg) three times a week.
  Interventions: Drug: ATRIPLA
- ATRIPLA one time a day. (Active Comparator): Atripla (600 mg/200 mg/245 mg) one time a day.
  Interventions: Drug: ATRIPLA

INTERVENTIONS:
Drug: ATRIPLA
  Other Names: efavirenz/emtricitabine/tenofovir disoproxil fumarate 600 mg/200; mg/245 mg

SUMMARY:
The main objective is to determine the feasibility of maintaining virologic suppression on standard plasma viral load by dose reduction of ATRIPLA ®.

DETAILED DESCRIPTION:
The main objective of this study is to determine the feasibility of maintaining virologic suppression on standard plasma viral load (limit of detection 37 copies / mL) of a dose reduction strategy of ATRIPLA ® once a day to three tablets per week in patients infected with HIV-1 with sustained suppression of plasma viral load standard for more than two years.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* HIV-1 infection, clinical stability, and treatment with ATRIPLA ® for the past two years.
* Standard plasma viral load below the limit of detection for at least 2 years.
* CD4 count above 350/mm3 at the time of the consideration for the study.
* Negative pregnancy test in women of childbearing age, and commitment acceptable contraceptive use for at least 2 weeks before day 1 and until at least 6 months after the last dose of study drug.
* Patients should be given written informed consent
* In the opinion of the investigator, be able to follow the design of the protocol visits

Exclusion Criteria:

* Patients who have experienced virologic failure prior to any antiretroviral regimen
* Evidence of previous mutations versus efavirenz, tenofovir and emtricitabine
* Use of any other chronic treatment plus ATRIPLA has been introduced in the 6 months prior to entry of the patient in the study
* Any contraindication to study drug
* Any condition not ensure proper adherence to the study at the discretion of the attending physician of the patient
* Uncontrolled preexisting psychiatric illness
* Any current sign of alcoholism or other drug use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2014-11-14 (Actual); Study Completion 2015-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Martinez, MD, Principal Investigator — Hospital Clínic i Provincial de Barcelona
Locations (1):
- Hospital Clinic i Provincial Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Guardo AC, Zarama A, Gonzalez T, Bargallo ME, Rojas J, Martinez E, Plana M, Sanchez-Palomino S. Effects on immune system and viral reservoir of a short-cycle antiretroviral therapy in virologically suppressed HIV-positive patients. AIDS. 2019 May 1;33(6):965-972. doi: 10.1097/QAD.0000000000002169. PMID 30946150
- [Derived] Rojas J, Blanco JL, Sanchez-Palomino S, Marcos MA, Guardo AC, Gonzalez-Cordon A, Lonca M, Tricas A, Rodriguez A, Romero A, Miro JM, Mallolas J, Gatell JM, Plana M, Martinez E. A maintenance 3-day-per-week schedule with the single tablet regimen efavirenz/emtricitabine/tenofovir disoproxil fumarate is effective and decreases sub-clinical toxicity. AIDS. 2018 Jul 31;32(12):1633-1641. doi: 10.1097/QAD.0000000000001843. PMID 29746294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 3 June 2013 and 30 May 2014 at Hospital Clínic of Barcelona.
Pre-assignment Details: 68 patients were assessed for eligibility, 61 underwent randomization and received at least one dose of study drugs. Seven patients were excluded because of refusal to participate (lack of time, n¼4; lack of interest, n¼1; fear of viral failure, n¼1) or evidence of illicit drug consumption (n¼1).
Groups:
- ATRIPLA Three Days a Week (3W): Atripla (600 mg/200 mg/245 mg) three days a week (Mondays, Wednesdays and Fridays).
- ATRIPLA One Time a Day (OD): Atripla (600 mg/200 mg/245 mg) one time a day.
Period: Overall Study
Arm/Group | ATRIPLA Three Days a Week (3W) | ATRIPLA One Time a Day (OD)
Started | 30 | 31
Completed | 30 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATRIPLA Three Days a Week (3W) | ATRIPLA One Time a Day (OD) | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47.8 [37.4 to 53.8] | 48.5 [38.1 to 58.3] | 48.2 [38.0 to 54.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 27 | 27 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 11 | 10 | 21
  Ethnicity: Caucasian | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Free of Treatment Failure (Noncompleter = Failure) at 24 Weeks.
Description: Treatment failure defined as any of the following possibilities occurring within the 24-week study framework: virological failure (confirmed plasma viral load 37 copies/ml), discontinuation of the antiretroviral therapy schedule irrespective of the reason, consent withdrawal, lost to follow-up, pregnancy, inability to comply with the study or any other reason that could make the doctor in charge consider the cessation of the study.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ATRIPLA Three Days a Week (3W) | ATRIPLA One Time a Day (OD)
Number analyzed (Participants) | 30 | 31
Participants
  Patients free of treatment failure | 30 | 31
  Patients with treatment failure | 0 | 0

2. Secondary Outcome: The Proportion of Patients With Ultrasensitive Viral Load (<1 Copy / mL) After 24 Weeks.
Time Frame: 24 weeks
Reporting Status: Not Posted

3. Secondary Outcome: The Change From Baseline to 24 Weeks in the Viral Reservoir in Peripheral Blood Mononuclear Cells
Time Frame: baseline and 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Immunological
Description: Changes from baseline to 24 weeks in the production of TRECs, the immunological profile of activation (CD38 and HLA-DR) and senescence (CD57 and CD28) in CD4 and CD8 lineages in the proportions of naive T cells effector and memory (CCR7 and CD45RA), and changes in the levels of apoptosis in vitro by staining with annexin V.
Time Frame: baseline and 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Changes in Plasma Levels of Efavirenz.
Time Frame: baseline and 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Changes in Sleep Quality (Pittsburgh Sleep Quality Index).
Time Frame: baseline and 6 months
Reporting Status: Not Posted

7. Secondary Outcome: General Safety (Report Adverse Events, Serious Adverse Events and Treatment Discontinuation Due to Adverse Events)
Time Frame: 24 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Changes in Plasma Levels of Vitamin D.
Time Frame: baseline and 6 months
Reporting Status: Not Posted

9. Secondary Outcome: Changes in Lipid Profile.
Time Frame: baseline and 6 months
Reporting Status: Not Posted

10. Secondary Outcome: Changes in Estimated Glomerular Filtration Rate.
Time Frame: baseline and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: AE/SAE definitions were consistent with ClinicalTrials.gov, but also included clinically significant lab abnormalities and events related to overdose, abuse, or withdrawal.
  AEs were collected systematically at baseline, weeks 12 and 24 in both arms, and at weeks 1, 2, 4, 6, and 8 in the 3-day/week arm. Grading used DAIDS Table v1.0 (Dec 2004; Clarified Aug 2009).
Arm/Group | ATRIPLA Three Days a Week (3W) | ATRIPLA One Time a Day (OD)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 13/30 | 11/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATRIPLA Three Days a Week (3W) (N=30) | ATRIPLA One Time a Day (OD) (N=31)
Mild, non-serious adverse events (General disorders) | 13 (13) | 11 (11) — All reported events were grade 1-2, not related to study drug

LIMITATIONS AND CAVEATS:
This was a single-center, open-label, pilot study with a small sample size (N=61) and short follow-up (24 weeks). The study was not powered to detect rare adverse events or long-term outcomes. No formal non-inferiority analysis was conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT01778413/Prot_SAP_000.pdf